CLINICAL TRIAL: NCT03269981
Title: A Phase III Prospective Randomized Study of Elective Regional Lymph Node Irradiation in Pathologic N1 Breast Cancer Patients Treated With Breast Conserving Surgery
Brief Title: Randomized Study of Elective Regional Lymph Node Irradiation in N1 Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Radiation Oncology Group (Unknown); Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2017-01-085-001
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasm
Keywords: Adjuvant radiotherapy; Lymphatic irradiation; Taxane; Anthracycline; Prospective study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole breast irradiation (Experimental): Post-lumpectomy radiotherapy to the whole breast alone.
  Interventions: Radiation: Whole breast irradiation
- Whole breast and nodal irradiation (Active Comparator): Post-lumpectomy radiotherapy to the whole breast and regional lymph node.
  Interventions: Radiation: Whole breast and nodal irradiation

INTERVENTIONS:
Radiation: Whole breast irradiation — Radiotherapy to the whole breast alone.
  Arms: Whole breast irradiation
Radiation: Whole breast and nodal irradiation — Radiotherapy to the whole breast and regional lymph nodes.
  Arms: Whole breast and nodal irradiation

SUMMARY:
This study evaluates the impact of elective regional lymph node irradiation on N1 breast cancer patients receiving post-lumpectomy radiotherapy and anthracycline plus taxane (AT)-based chemotherapy. We randomly assign patients having one to three metastatic lymph nodes (pN1) after breast-conserving surgery (BCS) and AT-based chemotherapy to undergo either whole-breast and regional nodal irradiation (WB+RNI group) or whole-breast irradiation alone (WBI group).

DETAILED DESCRIPTION:
Objective:

* Compare the effect of post-BCS WBI vs. WB+RNI on disease-free survival in pN1 breast cancer patients who received AT-based chemotherapy.
* Evaluate the impact of WBI or WB+RNI according to molecular subtype of tumor.
* Compare the treatment-related toxicities between the WBI and WB+RNI.
* Compare the patient's quality of life between the WBI and WB+RNI.

Outline: This is a a randomized, multi-center, phase III study. Patients are stratified according to molecular subtype of tumor (luminal A vs luminal vs luminal HER2 vs HER2-enriched vs basal-like), axillary lymph node management (sentinel lymph node biopsy [SLN] only vs axillary lymph node dissection+/- SLN) and participating institutions. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive WB+RNI.
* Arm II: Patients receive WBI alone.

Arm circumference and quality of life (EORTC QLQ-C30 & EORTC QLQ-BR23) are assessed within 2 weeks prior to randomization, during the last week of radiotherapy, at 3 months after completion of radiotherapy, and then annually thereafter for five years.

Patients are followed at 3 months after completion of radiotherapy and annually thereafter for seven years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive carcinoma of the breast.
* One to three positive axillary lymph nodes (pN1) proven in pathologic specimen.
* Prior breast-conserving surgery and post-operative adjuvant chemotherapy including taxane.
* Administering adjuvant hormonal therapy in cases with hormone receptor-positive tumor.
* Administering anti-HER2 therapy in cases with HER2-positive tumor.

Exclusion Criteria:

* Metastases in supraclavicular or internal mammary lymph nodes.
* Metastases in distant organs.
* Neoadjuvant chemotherapy or hormone therapy before surgery.
* Not receiving adjuvant anthracycline and taxane.
* Bilateral breast cancer
* Previous history of radiotherapy of the ipsilateral breast or supraclavicular lymph nodes.
* Prior history of other types of cancer, except thyroid cancer, carcinoma in situ of the cervix, or skin cancer.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 7 years
  Disease-free survival

SECONDARY OUTCOMES:
Disease-free survival according to molecular subtype | 5 years
  Disease-free survival according to molecular subtype
Treatment-related toxicity | 5 years
  acute and chronic toxicities
European Organization for Research and Treatment of Cancer (EORTC)-Quality of life. Questionnaire 30 (QLQ-C30) measurement | 5 years
  1 (Not at all) to 4 (Very much), 1 (Very poor) to 7 (Excellent). For functional and global quality of life scales, higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
EORTC Quality of Life Questionnaire - Breast Cancer Module (EORTC QLQ-BR23) measurement | 5 years
  1 (Not at all) to 4 (Very much). A higher score means more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided